CLINICAL TRIAL: NCT04023318
Title: A Novel Integrated Lifestyle Intervention to Reduce Obesity and Inflammation Among Emerging Adults
Brief Title: The BMI Project (Body, Mind, Inflammation)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18-14509; HM20015075 (Other: Virginia Commonwealth University IRB); NCI-2019-04792 (Other: National Cancer Institute)
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Overweight and Obesity; Chronic Inflammation
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Integrated Lifestyle Intervention (Experimental)
  Interventions: Behavioral: Integrated Lifestyle Intervention

INTERVENTIONS:
Behavioral: Integrated Lifestyle Intervention — This program is grounded in data demonstrating the dysregulation across multiple domains and considerable life stressors experienced by this population. The central hypothesis is that by simultaneously ameliorating psychological dysregulation and directly targeting proinflammatory behaviors, ILI operates on multiple proposed mediators of poor treatment outcomes in this population, thereby enhancing treatment outcomes. As such, the overall framework emphasizes integration of self-regulation as it applies to both psychological functioning and weight control. Content will highlight the interconnectedness of mood, stress, eating and exercise behaviors, and risk for inflammation and disease. Each treatment session will present a combination of behavioral and psychological content, representing a truly integrated approach. Participants will meet for 75-minute group sessions weekly for months 1-2, followed by bi-weekly groups in months 3-4, for a total of 12 groups.

SUMMARY:
Obesity and chronic inflammation influence the development and progression of many types of cancer. These conditions share several of the same causes, including physical inactivity, poor nutrition, stress, and insufficient sleep. Emerging adulthood (ages 18-25) represents an important developmental period in which to address behaviors and psychological variables that affect both weight status and inflammation. At least 40% of emerging adults have overweight/obesity, and this transition from adolescence to early adulthood is associated with significant increases in fast food consumption, decreases in physical activity, unpredictable sleep schedules, and alarmingly high rates of depression and perceived stress.

Despite this high risk for obesity, very few weight loss interventions are designed specifically for emerging adults. Preliminary findings from weight loss interventions targeting this population have shown some promise, but generally produce modest outcomes with less consistent effects than programs in older adults. Depression and stress have been found to interfere with weight loss among emerging adults, and may be in part responsible for poorer outcomes. This proposal will develop and test an Integrated Lifestyle Intervention (ILI) that comprehensively addresses both psychological distress and traditional weight management targets. This novel approach has not been tested before and has the potential not only to enhance weight loss outcomes in this high risk population, but also to produce reductions in markers of inflammation beyond those achievable by weight loss alone.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 25 years
* Body Mass Index between 25 and 45 kg/m2

Exclusion Criteria:

* Currently pregnant or lactating; pregnancy in the last 6 months or plans to become pregnant in the next 6 months
* Type 1 or type 2 diabetes
* Any uncontrolled medical conditions that could make it unsafe to participate in unsupervised exercise
* Medical conditions associated with chronic inflammation
* Inability to read, understand and speak English

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Number of sessions attended throughout the intervention period | 4 months
  Attendance at in-person treatment sessions is one critical metric for demonstrating feasibility and will be tracked throughout the intervention period.
Number of days self-monitoring weight in LoseIt | 4 months
  Self-monitoring of weight is a critical metric for demonstrating feasibility and will be tracked throughout the intervention period.
Number of days self-monitoring weight-related behaviors in LoseIt | 4 months
  Self-monitoring of weight-related behaviors (e.g., diet and physical activity) is a critical metric for demonstrating feasibility and will be tracked throughout the intervention period.

SECONDARY OUTCOMES:
Change in diet | Baseline and 4 months
  Dietary change will be assessed using the Diet History Questionnaire III (DHQ-III), a 166-item adaptive questionnaire developed by NCI which maps on to dietary intervention targets (e.g., saturated fat, alcohol, sugar, fiber, sodium), as well as a measure of overall diet.
Change in physical activity | Baseline and 4 months
  Participants will report their physical activity using the 6-item Paffenbarger Physical Activity Questionnaire, which yields estimates of minutes spent in moderate-to-vigorous physical activity.
Change in sleep | Baseline and 4 months
  The EARLY Trials Common Elements Sleep Questionnaire (8 items) will be administered that asks about duration of sleep and problems encountered during sleep (e.g. snoring).
Percent Weight Change | Baseline and 4 months
  Weight will be measured in light clothes, without shoes, on calibrated Tanita BWB-800S scales. Percent change of initial body weight will be calculated using baseline and 4 month weights.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica LaRose, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT04023318/ICF_000.pdf